CLINICAL TRIAL: NCT06426238
Title: Comparison of Self-reported and Experimental Pain Outcomes Between Clear Aligners and Fixed Appliances in Patients Undergoing Orthodontic Treatment
Brief Title: Self-reported and Experimental Pain in Patients Undergoing Orthodontic Treatment
Status: Completed | Type: Observational
Sponsor: Midwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: CIRB_23010
Record Dates: First submitted 2024-05-07; First posted 2024-05-23 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Pain
Keywords: Pressure pain threshold; Clear aligners; Orthodontic appliance; Adolescents; Self-reported pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pressure Pain Threshold (PPT) is defined as the minimum force applied to an area that is perceived as pain. PPT is considered an objective measurement tool to assess pain levels. Studies have assessed the difference in pain levels between clear aligners and fixed appliances using subjective pain scales. No study has utilized PPT to evaluate the difference in pain between aligners and fixed braces at different time points. This study will aim to compare the self- reported and experimental pain perception between the clear aligner and fixed appliance therapies during the phase of crown alignment and to assess how long pain is perceived in the following five days from the adjustment of the appliance.

ELIGIBILITY:
Inclusion Criteria:

* consecutive consented patients (> 14 years old) beginning an orthodontic treatment on both arches, either with aligners or fixed appliance at the Midwestern University, Multidisciplinary Clinic;
* patients in possession of an email address and Internet connection.

Exclusion Criteria:

* patients with generalized systemic conditions known to affect the overall body pain and pressure pain threshold assessment (e.g., fibromyalgia, autoimmune conditions such as multiple sclerosis, rheumatoid arthritis),
* untreated dental caries.

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients starting an orthodontic treatment (clear aligners or fixed braces) at the Multispecialty Clinic of Midwestern University
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Self-reported pain intensity | At three timepoints through study completion: at baseline, at 4-6 weeks, and at 8-12 weeks
  Self-reported pain will be assessed using a Visual Analogue Scale with anchors from 0 (=no pain) to 10 (=worst imaginable pain)
Pressure Pain Threshold | At three timepoints through study completion: at baseline, at 4-6 weeks, and at 8-12 weeks
  Pressure Pain Threshold will be measured through an algometer on masseter and temporals muscles

SECONDARY OUTCOMES:
Anxiety and depression symptoms | At two timepoints through study completion: at baseline, and at 8-12 weeks
  Self-perceived anxiety and depression measured through the Patient Health Questionnaire, PHQ-4 (from 0 to 12, with higher score identifying higher anxiety and depression)
Pain catastrophizing | At two timepoints through study completion: at baseline, and at 8-12 weeks
  Self-reported pain catastrophizing measured trough Pain Catastrophizing Scale, PCS (from 0 to 52, with values >30 identifying clinically meaningful pain catastrophizing)
Past pain experience | At T0: Baseline (pre-intervention)
  Semi-structural interview through questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Midwestern University, Downers Grove, Illinois, United States